CLINICAL TRIAL: NCT03163043
Title: Evaluation of Protein Requirements in Active Children
Brief Title: Protein Requirements for Active Children
Acronym: IAAO-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Moore (Other)
Collaborators: Ajinomoto Co., Inc. (Industry)
Responsible Party: Sponsor-Investigator, Daniel Moore, Dr. Daniel Moore, Assistant Professor, University of Toronto
Organization: University of Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IAAO-C
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Increased Metabolic Requirement; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active, Male and Female Children (Experimental): Participants will receive different levels of amino acid intakes, varying from 0.2-2.67 g/kg/d
  Interventions: Dietary Supplement: Amino Acid Intake

INTERVENTIONS:
Dietary Supplement: Amino Acid Intake — Amino acid intakes will be varied at 0.2-2.67 g/kg/d

SUMMARY:
Nutritional requirements for dietary amino acids in children have traditionally been determined utilizing the nitrogen balance technique, which is prone to underestimating protein requirements. As a result, there is a need to re-evaluate recommendations in order to characterize how dietary amino acid needs may be modulated by physical activity in healthy, active children. The purpose of this study is to measure the protein requirement in children (boys and girls) using the IAAO technique in the presence of a variable intensity exercise stimulus. It is hypothesized that the present study will deem current amino acid requirements to be underestimates of appropriate amino acid requirements for this population.

DETAILED DESCRIPTION:
Provided energy needs are met, the adequate ingestion of dietary amino acids is the most critical nutritional factor to support the optimal remodeling and deposition of lean body mass in individuals of all ages, including active youth. Despite the fact that the most consistent and rapid growth velocities outside of infancy occur during childhood and adolescence, respectively, there is a paucity of research into the fundamental questions of how exercise and nutrition (i.e. dietary amino acid ingestion) enhance protein turnover in these key demographics. Of primary importance is the impact exercise has on the nutritional requirement for dietary amino acids in concurrently growing youth. This lack of dedicated research represents a significant knowledge gap for a large segment of the world's population. Nutritional requirements for dietary amino acids in young adults has traditionally been determined utilizing the antiquated and often erroneous nitrogen balance technique, which makes it difficult to adequately define the protein needs of this population, let alone those of children. In addition, nitrogen balance requires a prolonged adaptation period, which exposes subjects to deficient intakes for 7-10 days, making it unsuitable for use in vulnerable populations like children. As a result, there is a need to establish (in the case of children) recommendations utilizing advanced stable isotope methodology in order to characterize how dietary amino acid needs may be affected by physical activity over the critical early years of development.

Studies using the minimally invasive indicator amino acid oxidation (IAAO) technique have suggested that protein requirements in young men and children are at least 50% higher than WHO/FAO guidelines based on nitrogen balance data.

The present study will use, for the first time in active children, the gold-standard IAAO technique to achieve two major objectives: i) to determine the impact of high levels of physical activity on protein requirements in active, growing children, and; ii) to determine whether exercise in adolescence, previously determined in a separate study, alters protein requirements relative to similarly active children.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, active children who regularly participates in moderate to vigorous physical activity 5 times a week for a minimum of 1 hour.
* Biological age less than or equal to -1.0 years from Peak Height Velocity (PHV), determined by the ratio of standing to sitting height
* An age and sex-specific minimum performance level on the Beep Test

Exclusion Criteria:

* Inability to meet health and physical activity guidelines according to the PAR-Q+ and Physical Activity Questionnaire
* Inability to adhere to any of the protocol guidelines (i.e., caffeine consumption)
* Biological age greater than -1.0 years from PHV

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2016-10-22 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
13CO2 ([13]Carbon Dioxide) Excretion (µmol/kg/h) | 4 hours/study day

SECONDARY OUTCOMES:
[13C]Phenylalanine Oxidation (µmol/kg/h) | 4 hours/study day

CONTACTS AND LOCATIONS:
Locations (1):
- Goldring Centre For High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No